CLINICAL TRIAL: NCT03770715
Title: Sleep Apnea After Extubation
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jaeyoung Cho, Assistant Professor, Seoul National University Hospital
Other Study IDs: 1802051921
Record Dates: First submitted 2018-12-07; First posted 2018-12-10 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Sleep Apnea
Keywords: Sleep Apnea; Respiratory polygraphy; Extubation
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Respiratory polygraphy — The respiratory polygraphy consisted of continuous polygraphical recordings for a whole night from 22:00 h to 07:00 h with standardised equipment

SUMMARY:
Sleep apnea is common after extubation, approximately 71%, and is independently associated with hypertension and metabolic disease contributing to increased morbidity and mortality. Respiratory polygraphy is a simpler alternative to in-laboratory polysomnography for the management of more symptomatic patients with obstructive sleep apnea.

The aim of this study is to evaluate the prevalence of sleep apnea after extubation by respiratory polygraphy.

ELIGIBILITY:
Inclusion Criteria:

* patients after extubation

Exclusion Criteria:

* pregnant
* non-consciousness
* received continuous positive airway pressure (CPAP)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary referral hospital
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2018-08-17 (Actual); Primary Completion 2019-05-24 (Actual); Study Completion 2019-12-02 (Actual)

PRIMARY OUTCOMES:
Prevalence of sleep apnea after exutbation | during first to second night following extubation

CONTACTS AND LOCATIONS:
Overall Officials: Jaeyoung Cho, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea